CLINICAL TRIAL: NCT04847102
Title: A Global, Multi-center, Randomized, Double-Blind, Placebo-controlled, Phase III Clinical Study to Evaluate the Protective Efficacy, Safety and Immunogenicity of SARS-CoV-2 Messenger Ribonucleic Acid (mRNA) Vaccine in Population Aged 18 Years and Older
Brief Title: A Phase III Clinical Study of a SARS-CoV-2 Messenger Ribonucleic Acid (mRNA) Vaccine Candidate Against COVID-19 in Population Aged 18 Years and Above
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walvax Biotechnology Co., Ltd. (Industry)
Collaborators: Abogen Biosciences Co. Ltd. (Industry); Yuxi Walvax Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: ARCoV-005
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: SARS-CoV-2 mRNA vaccine; Efficacy; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Biological: SARS-CoV-2 mRNA Vaccine; Biological: Placebo
- Control group (Placebo Comparator)
  Interventions: Biological: SARS-CoV-2 mRNA Vaccine; Biological: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 mRNA Vaccine — The SARS-CoV-2 mRNA Vaccine is formulated by encapsulating the mRNA, which encodes the receptor-binding domain (RBD) of spike glycoprotein (S protein) of SARS-CoV-2 and is transcribed in-vitro by the corresponding DNA template, in lipid nanoparticles (LNPs). This vaccine is presented as a white to off-white dispersion for injection.
  Active substances: mRNA encoding the RBD of the S protein of SARS-CoV-2.
  The vaccine is supplied in single-dose pre-filled syringe with 0.5 mL dispersion for intramuscular injection. Each dose (0.5 mL) of the vaccine contains:
  15 μg of mRNA encoding the RBD of the spike glycoprotein (S protein) of SARS-CoV-2, 0.339 mg of total lipids (including lipid 9001, cholesterol, DSPC, DMG-PEG2000).
Biological: Placebo — 0.9% sodium chloride solution, 0.5 mL/vial

SUMMARY:
Approximately 28,000 subjects will be enrolled in this trial. Eligible subjects will be stratified by age (<60 years of age and ≥60 years of age, the proportion of elderly people ≥60 years old is planned to be ≥25%) and randomly assigned into the study group and the control group at a ratio of 1:1 (14,000 in each group) to be intramuscularly administered with the investigational vaccine or placebo in a 2-dose regimen at an interval of 28 days. The experimental vaccines will be cross-vaccinated after available data of the investigational vaccine show that expected efficacy and good safety have been achieved (i.e., subjects in the study group will be vaccinated with placebo and those in the control group will be vaccinated with the investigational vaccine in the same schedule as stated above ). After the completion of the second dose for crossover vaccination, subjects will be followed up for 12 months for safety observation. An immunogenicity subgroup (n≥3000) and a reactogenicity subgroup (n≥6000) will also be included in this trial to evaluate the humoral immunity induced by the investigational vaccine and the solicited adverse events observed within 7 days post immunization. All enrolled subjects will be followed up for the evaluation of protective efficacy as well, which will be primarily characterized by the incidence rate (person-year) of COVID-19 cases collected from 14 days after complete series. Adverse events will be collected over 0-28 days after each vaccination and serious adverse events will be collected from Dose 1 through 12 months post complete series.

ELIGIBILITY:
Inclusion Criteria:

Subjects included in this trial must meet all of the following inclusion criteria:

1. Adults aged 18 and above (both males and females are required);
2. Individuals who are able to understand the contents listed in the informed consent form and the procedure of this clinical trial; are able to sign the informed consent form voluntarily;
3. Individuals who are able to communicate well with the investigator and has the ability to understand and comply with the requirements of the clinical trial;
4. Individuals who are at risk of SARS-CoV-2 infection or are exposed to COVID-19 due to regional, occupational, activity and environmental factors;
5. For female participants of childbearing potential, effective contraception should be used within 2 weeks prior to participation in this study and the pregnancy test results is required to be negative (those with amenorrhea of at least 1 year or surgical sterilization verified by medical records could be exempted from the pregnancy test). Participants should voluntarily agree to continue using at least one effective methods of contraception for 12 months after complete series (effective methods include oral contraceptives, injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).
6. Healthy individuals with verified medical history: individuals who are in a stable condition and whose current diseases will not worsen for at least 3 months prior to enrollment to this study.

Exclusion Criteria:

Exclusion criteria for first dose vaccination

Subjects who meet any of the following exclusion criteria shall not be enrolled:

1. Individuals with a history of SARS-CoV-2 infection or use of any preventive products for COVID-19 (e.g., a history of any SARS-CoV-2 vaccines that have or have not been marketed);
2. Individuals with SARS-CoV-2 etiological testing (RT-PCR Assay) (individuals with serological testing showing positive IgG and/or IgM antibodies may be enrolled);
3. Individuals with a previous history of severe acute respiratory syndrome (SARS), middle east respiratory syndrome (MERS) and other human coronavirus infections or diseases;
4. Individuals who have fever within 72 hours prior to Dose 1 in this trial (oral temperature ≥38°C);
5. Pregnant (e.g., positive pregnancy test) or lactating females;
6. Individuals who have plan of pregnancy or interruption of effective contraceptive methods within 3 months after the second cross-vaccination in this study;
7. Personnel of the study site or the sponsor;
8. Individuals with prior history of allergic reaction or anaphylaxis to any vaccine or drug, e.g., hypersensitivity, urticaria, serious eczema, dyspnea, laryngeal edema, and angioedema etc.;
9. Individuals who have been vaccinated with any vaccine other than the investigational vaccine used in this clinical trial from 28 days prior to Dose 1 to 28 days after Dose 2;
10. Individuals who have participated in or plan to participate in other drug clinical trials form 28 days prior to Dose 1 to 12 months after Dose 4 (the second dose of cross-vaccination) in this study;
11. Individuals who have hereditary hemorrhagic tendency or coagulation dysfunction (e.g., cytokine defects, coagulation disorders or platelet disorder), or a history of significant bleeding, or a history of injury caused by intramuscular injection or venipuncture;
12. Individuals who are confirmed for diseases affecting immune system function, including cancer (except skin basal cell carcinoma), congenital or acquired immunodeficiency (e.g., infection with human immunodeficiency virus (HIV)), and uncontrolled autoimmune disease, based on known history or diagnosis;
13. Individuals who have asplenia or functional asplenia;
14. Individuals with long-term use (continuous use ≥14 days) of immunosuppressants or other immunomodulatory drugs (e.g., corticosteroids: prednisone or similar drugs) within 6 months prior to Dose 1. Drugs for topical use (e.g., ointment, eye drops, inhalants or nasal spray) are allowed in this study, and the topical medications should not exceed the recommended dose in the labels for use or induce any signs of systemic exposure;
15. Individuals who have received immunoglobulin and/or blood products within 3 months prior to Dose 1;
16. Individuals who are suspected or known to have alcohol dependency problems or drug abuse that may affect safety evaluation or subject's compliance;
17. Individuals who plan to permanently relocate from the local area before the completion of the study or leave the local area for long periods during the study visits;
18. Other circumstances considered by the investigator as inappropriate to participate in the study.

Criteria for Postponement of the Subsequent Doses:

If the subjects have any of the followings prior to the subsequent doses, vaccination will be postponed. During the same immunization schedule, the second dose of vaccine will be administered at the 28th day after the first vaccination, with a time window of +5 days:

1. Fever within 72 hours prior to the subsequent doses (oral temperature ≥38°C, probability of SARS-CoV-2 infection shall be excluded);
2. In case of acute diseases prior to the subsequent doses, the investigator shall exclude the probability of SARS-CoV-2 infection and evaluate the likelihood of short-term recovery for the diseases;

Exclusion Criteria for the Subsequent Doses:

If the subject has any of the followings prior to the subsequent doses, the vaccination shall be terminated for the subject while other study procedures could be continued at the discretion of the investigators:

1. Female subjects of childbearing potential who have positive pregnancy test results;
2. Subjects who have a serious allergic reaction or serious adverse event causally related to vaccination after previous vaccination;
3. Other circumstances considered by the investigator as inappropriate to receive the subsequent doses of the vaccine.

Criteria for Withdrawal from the Study

1. Subjects experience disability, life-threatening adverse events or serious adverse events and have to prematurely withdraw from this study due to treatment or other reasons.
2. Subjects are placed at safety risks by their health conditions which prevent them from continuing to participate in this study.
3. Female subjects become pregnant during the study (if at least one dose has been administered, the subject is not required to withdraw from this study but should not receive the subsequent doses. Moreover, subsequent observation and follow-up visits should be continued);
4. Subjects actively request to withdraw from the study;
5. Subjects are considered unsuitable for continuing to participate in this study at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28000 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint as measured by the incidence rate (person-year) of COVID-19 cases | From 14 days after complete series
  The incidence rate (person-year) of COVID-19 cases collected from 14 days after complete series in subjects aged 18 years and above.
Primary safety endpoint as measured by the incidence rates of adverse events | Within 28 days post each vaccination
  Incidence rates of adverse events observed for all subjects within 28 days post each vaccination;
Primary safety endpoint as measured by the incidence rates of serious adverse events | At 7 days post each vaccination
  Incidence rates of solicited adverse events observed for subjects included in the reactogenicity subgroup within 30 minutes and at 7 days post each vaccination.

SECONDARY OUTCOMES:
Secondary efficacy endpoint as measured by the incidence rate (person-year) of severe and critical COVID-19 cases | From 14 days after complete series
  The incidence rate (person-year) of severe and critical COVID-19 cases collected from 14 days after complete series in subjects aged 18 years and above;
Secondary efficacy endpoint as measured by the incidence rate (person-year) of COVID-19 cases resulting in deaths | From 14 days after complete series
  The incidence rate (person-year) of COVID-19 cases resulting in deaths collected from 14 days after complete series in subjects aged 18 years and above;
Secondary efficacy endpoint as measured by the incidence rate (person-year) of COVID-19 cases post 1 dose of vaccination | From 14 days after Dose 1
  The incidence rate (person-year) of COVID-19 cases collected from 14 days collected after Dose 1 in subjects aged 18 years and above who fail to be administered with Dose 2 for personal reasons.
Secondary safety endpoint as measured by the incidence rate of serious adverse events | From Dose 1 through 12 months after complete series
  Incidence rates of serious adverse events observed for all subjects from Dose 1 through 12 months after complete series.

CONTACTS AND LOCATIONS:
Locations (12):
- Indonesia (5):
  - Persahabatan Hospital, Jakarta
  - Puskesmas Duren Sawit, Jakarta
  - Puskesmas Kalideres, Jakarta
  - Puskesmas Kebayoran Lama, Jakarta
  - Puskesmas Pulogadung, Jakarta
- Mexico (7):
  - Centro de Investigación Clínica del Pacifico S.A. de C.V. (CICPA), Acapulco
  - Centro de Investigación y Avances Médicos Especializados (CIAME), Cancún
  - Centro de Especialidades Médicas Aplicadas, Mexico City
  - Instituto Nacional de Pediatría (INP), Mexico City
  - Oaxaca site management organization (OSMO), Oaxaca City
  - Asociación Mexicana para la investigación clínica, A.C. (AMIC), Pachuca
  - Oncológico Potosino, San Luis Potosí City

REFERENCES:
- [Derived] Liu X, Li Y, Wang Z, Cao S, Huang W, Yuan L, Huang YJ, Zheng Y, Chen J, Ying B, Xiang Z, Shi J, Zhao J, Huang Z, Qin CF. Safety and superior immunogenicity of heterologous boosting with an RBD-based SARS-CoV-2 mRNA vaccine in Chinese adults. Cell Res. 2022 Aug;32(8):777-780. doi: 10.1038/s41422-022-00681-3. Epub 2022 Jun 14. No abstract available. PMID 35701541
- [Derived] Zhang NN, Zhang RR, Zhang YF, Ji K, Xiong XC, Qin QS, Gao P, Lu XS, Zhou HY, Song HF, Ying B, Qin CF. Rapid development of an updated mRNA vaccine against the SARS-CoV-2 Omicron variant. Cell Res. 2022 Apr;32(4):401-403. doi: 10.1038/s41422-022-00626-w. Epub 2022 Feb 14. No abstract available. PMID 35165421